CLINICAL TRIAL: NCT00743197
Title: Women With Chest Pain and Normal Coronary Arteries Study: A Randomized Study of Medical Treatment and Therapeutic Lifestyle Changes
Brief Title: Women With Chest Pain and Normal Coronary Arteries Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to departure of PI from institution.
Sponsor: Northwestern University (Other)
Collaborators: Astellas Pharma US, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: AB-08-002
Record Dates: First submitted 2008-08-26; First posted 2008-08-28 (Estimated); Results first posted 2011-11-23 (Estimated); Last update posted 2023-12-12 (Actual); Status verified 2023-11

CONDITIONS: Chest Pain
Keywords: coronary artery disease (CAD); chest pain; myocardial ischemia; endothelial function
MeSH Terms: conditions — Chest Pain; Coronary Artery Disease; Myocardial Ischemia | interventions — Aspirin; Lisinopril; Simvastatin; Omacor; Fish Oils; Docosahexaenoic Acids

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual Care Group (No Intervention): USUAL CARE GROUP-therapy in this group will be no dictated medical therapy, but usual care, as dictated by their referring physician.
- Medical Treatment Group (Active Comparator): TREATMENT GROUP-therapy in this group will be conventional treatment for CAD but targeting endothelial function, which will include aspirin, ACE-inhibitor and statin therapy, and therapeutic lifestyle changes.
  Interventions: Drug: Aspirin; Drug: Lisinopril; Drug: Simvastatin; Drug: Lovaza; Behavioral: Therapeutic Lifestyle Changes

INTERVENTIONS:
Drug: Aspirin — Aspirin 81 mg daily
  Arms: Medical Treatment Group
Drug: Lisinopril — Lisinopril 10 mg every night
  Arms: Medical Treatment Group
Drug: Simvastatin — Simvastatin 20 mg every night
  Other Names: Zocor
  Arms: Medical Treatment Group
Drug: Lovaza — Lovaza 1 gram daily
  Other Names: Fish Oil, Omega-3
  Arms: Medical Treatment Group
Behavioral: Therapeutic Lifestyle Changes — Therapeutic lifestyle changes will be initiated with the assistance of a dietician, including diet counseling, exercise recommendation, and weight maintenance/weight loss.
  Arms: Medical Treatment Group

SUMMARY:
The purpose of this study is to compare the effectiveness of standard medical therapy versus usual care in women with chest pain, coronary endothelial dysfunction and unblocked coronary arteries.

Coronary endothelial dysfunction (CED) is a condition in which the layers of cells around the heart do not function properly and is believed to be key factor in the development of atherosclerosis (fat deposits in arteries). In addition, CED is associated with an increased risk for future cardiovascular events, such as heart attack and stroke.

A coronary angiogram allows physicians to see if any of the arteries in the heart are blocked, usually by fatty plaque. In many instances, angiograms in women experiencing chest pain do not show evidence of coronary disease (free of significant plaque build-up). Currently, there is no standard of care treatment plan for patients with normal coronary arteries, despite symptoms of chest pain, and as a result these patients may not receive medical treatment. However, these women often return to their physicians more than once with chest pain and go through a similar battery of tests.

DETAILED DESCRIPTION:
Endothelial function testing will be performed on women without significant coronary disease in order to help identify women who may be likely to develop coronary artery disease (CAD) and who would benefit from aggressive lifestyle (dietary counseling, exercise) or medical (treatment with aspirin and cholesterol and blood pressure lowering medications) interventions.

ELIGIBILITY:
Inclusion Criteria:

1. Female gender
2. Age 30 or greater
3. Present with symptoms suggestive of Angina (Typical or "Atypical")
4. Abnormal myocardial perfusion scan
5. Referred for angiography
6. Normal (0% stenosis) versus Nonobstructive coronary artery disease (CAD) (<50% stenosis)
7. Evidence of endothelial dysfunction.

Exclusion Criteria:

1. Coronary vasospasm known or documented in cardiac catheterization
2. Obstructive CAD (greater than 50% stenosis) known or documented in cardiac catheterization
3. Pregnancy
4. Established CAD, history of revascularization with percutaneous transluminal coronary angioplasty (PTCA)/stent or coronary artery bypass graft (CABG)
5. Contraindications to magnetic resonance imaging (MRI)
6. Cardiac catheterization for valvular disease
7. Cardiac catheterization for heart failure assessment/biopsy
8. Known congestive heart failure (CHF)/hypertrophic obstructive cardiomyopathy (HOCM)/dilated cardiomyopathy (DCM)
9. Acute Renal Failure
10. Chronic renal failure (estimated glomerular filtration rare (eGFR) <30 ml/min/1.73m^2) or on hemodialysis
11. Known single kidney
12. History of peptic ulcer disease, known gastrointestinal bleed, known contraindication to aspirin
13. Known contraindication to statin
14. Known contraindication to adenosine (asthma, high degree atrial ventricular (AV) block)

Ages: 30 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Martha Gulati, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Usual Care Group | Medical Treatment Group
Started | 1 | 2
Completed | 0 | 0
Not Completed | 1 | 2
Not completed — Study terminated due to departure of PI. | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Usual Care Group | Medical Treatment Group | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Effectiveness of Therapy Compared to Usual Care, in Those Women With Chest Pain (CP), Reversible Ischemia by Stress Testing and Nonobstructive Coronary Artery Disease (CAD) by Angiography Who Are Found to Have Coronary Endothelial Dysfunction (CED).
Description: The purpose of this study is to compare the effectiveness of standard medical therapy versus usual care in women with chest pain (CP), coronary endothelial dysfunction (CED) and unblocked coronary arteries. CED is a condition in which the layers of cells around the heart do not function properly and is believed to be a key factor in the development of atherosclerosis (fat deposits in arteries). In addition, CED is associated with an increased risk for suture cardiovascular events, such as heart attack and stroke.
Time Frame: 1 year
Population: no analyses were conducted due to PI's departure from institution;all work including analyses ceased upon departure-the study was not transferred with the PI. In addition, study end points were based on changes between groups (treatment vs. usual care)at 12-mo follow up for both groups- none of the enrolled subjects completed the month 12 visit.
Arm/Group | Usual Care Group | Medical Treatment Group
Number analyzed (Participants) | 0 | 0
Statistical Analysis 1: Comparison: Usual Care Group vs Medical Treatment Group; 0; Test type: Non-Inferiority or Equivalence — 0; 0; Other = 0, Standard Deviation 0

ADVERSE EVENTS:
Arm/Group | Usual Care Group | Medical Treatment Group
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/1 | 0/2

LIMITATIONS AND CAVEATS:
Study terminated due to departure of PI; all work including analyses ceased upon departure.In addition,study end points were based on changes b/w groups treatment vs. usual care) at 12 mo follow up- none of the subjects completed the Mo 12 visit.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes